CLINICAL TRIAL: NCT02264548
Title: A Phase I Study Evaluating the Integration of Hypofractionated Renal Ablative Radiotherapy in the Setting of Metastatic Renal Cell Carcinoma
Brief Title: A Phase I Evaluating Integration of HypofractionatedStudy Renal Ablative Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Belal Ahmad, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renal Ablation
Record Dates: First submitted 2014-07-22; First posted 2014-10-15 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Radiation: Radio-Ablation
  Interventions: Radiation: Radio-Ablation

INTERVENTIONS:
Radiation: Radio-Ablation — Level I 20Gy/5 Level II 25Gy/5 Level III 30Gy/5 Level IV 35Gy/5 Level V 40Gy/5

SUMMARY:
* evaluate the safety and toxicity profile of renal radio-ablation in the setting of metastatic renal cell carcinoma.
* to assess renal function post radio-ablation
* Primary and metastatic tumour response to radio-ablation

DETAILED DESCRIPTION:
A dose limiting toxicity (DLT) will be defined as any grade 3, 4 or 5 toxicity event that is considered to be definitely, probably or possibility related to the protocol radiation therapy. Patients that cannot complete protocol therapy due to acute radiation side-effects will also be considered to be a DLT. The general (non-exhausive) list of organ based toxicity that could be related to this type of radiation therapy include toxicity to the liver, kidney, bowel, spinal cord, and pancreas. Side-effects that are exclusively due to TKI targeted therapy are not considered to be DLT in this protocol.

Three patients will be recruited for the first cohort of the trial. These patients will have the PTV prescribed a dose of 25 Gray to be given in 5 daily fractions over a period of one week (first treatment to start on a Wednesday or Thursday, with planned treatment on successive business days). All therapy should be delivered within 10 business days including any treatment breaks for acute toxicity. After 3 patients have been seen at the 4 week follow up visit, CTCAE version three will be noted. If precisely 1 patient has a DLT, then an additional 3 patients will be recruited to the same cohort and given the same treatment. If no patient has DLT, then a new cohort of 3 patients will be treated to an increased dose of 30 Gray in 5 fractions. Similar criteria will dictate whether the trial ends, or continues with the next cohort being treated to a dose of 35 Gray in 5 daily fractions. There will be a maximum of 4 cohorts (25Gy, 30Gy, 35Gy, and 40Gy) in this study assuming no early DLT issues, each containing 3 or 6 patients. Allowance for a -1 cohort arm of 20 Gy in 5 fractions is made in this protocol for early DLT issues. The diagram below displays the schema in more detail.

Any patient that does not complete protocol therapy due to toxicity issues or is unavailable for the 4-week toxicity assessment is considered to be non-evaluable. These patients will need to be replaced in terms of study accrual. Patients are not to be given TKI therapy during the 4 week window post-RT in order to allow for proper evaluation of the RT intervention; however, the treating oncologist ultimately can override this if it is in the best medical interest of the patient (e.g. progressive and symptomatic systemic disease)

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria

* Patients must have histologically confirmed carcinoma of the kidney
* Patients must be able to tolerate extended treatment time 30 minutes for MVCT and treatment delivery) for radiation on the tomotherapy unit
* Patients must have confirmed metastatic disease, nodal or locally advanced disease either by biopsy or imaging
* Informed consent performed and documented
* Patients must have one of a) unresectable local disease, b) be medically inoperable, or c) chosen against having a local surgical treatment
* Age ≥ 18
* Patients previously received any targeted therapy or immunotherapy for RCC, are also eligible. Patients must be off these agents for a minimum of 2 weeks prior to radiation therapy to be eligible

Exclusion Criteria:

* Patients without an adequate functioning contralateral kidney as seen on renal perfusion scan (>40% of total renal flow)
* Patients with poor baseline renal function, represented by a creatinine clearance < 50 mL/minute based on the Cockcroft-Gault approximation method
* Patients with a creatinine clearance < 50 ml/minute are still eligible if the ipsilateral kidney has <25% of the total renal flow on a renal perfusion scan.

еCCr =140 - (Age) × Mass (in kilograms) × constant Serum creatinine ( in µmol/L) constant = male is 1.23, women is 1.04)

* Previous abdominal radiotherapy
* Bilateral RCC
* Diagnosis of transitional cell carcinoma, squamous cell carcinoma, or a non epithelial cancer of the kidney
* Diagnosis of any other malignancy in previous 5 years, excluding non-melanoma skin cancer -Known active malignancy other than RCC, excluding non-melanoma skin cancer
* Estimated (by treating radiation oncologist) life expectancy of less than 8 weeks
* Pregnant or breast-feeding women
* Concurrent illness in addition to RCC that would make radiotherapy delivery unduly challenging, including but not limited to, severe congestive heart failure or other cardiorespiratory conditions, severe neuromuscular disorders, ongoing or active infections, and psychiatric illness
* Medical conditions for which radiation is contraindicated, including but not limited to, scleroderma, systemic lupus erythematosus and ataxia teleangiectasia - Patients with excessive kidney motion on pre-planning 4D-CT scan that would prevent safe delivery of radiotherapy with gated or non-gated techniques
* Patients taking concurrent medication that can interfere with the safe delivery of radiation (e.g. radiosensitizers)
* Urology opinion recommends partial nephrectomy as cytoreductive atment --Expected TKI therapy to be initiated during initial 2 weeks completion of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-07; Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
evaluate the safety/toxicity profile of renal radio-ablation in the setting of metastatic RCC | After 3 patients have been seen at the 4 week follow up visit,
  toxicity will be assessed using CTCAE v3

SECONDARY OUTCOMES:
Renal Function post renal radio-ablation | 4,8,12 wk and every 6months x 5yr
  BUN, Creatinine

OTHER OUTCOMES:
Tumour Response | 4,8,12 wk and every 6 months x5yr.
  CT abdomen evaluting primary disease using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Belal Ahmad, MD FRCPC, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program of the Laswon Research Health Institue, London, Ontario, Canada

REFERENCES:
- [Derived] Correa RJM, Ahmad B, Warner A, Johnson C, MacKenzie MJ, Pautler SE, Bauman GS, Rodrigues GB, Louie AV. A prospective phase I dose-escalation trial of stereotactic ablative radiotherapy (SABR) as an alternative to cytoreductive nephrectomy for inoperable patients with metastatic renal cell carcinoma. Radiat Oncol. 2018 Mar 20;13(1):47. doi: 10.1186/s13014-018-0992-3. PMID 29558966
- [Derived] Correa RJM, Rodrigues GB, Chen H, Warner A, Ahmad B, Louie AV. Stereotactic Ablative Radiotherapy (SABR) for Large Renal Tumors: A Retrospective Case Series Evaluating Clinical Outcomes, Toxicity, and Technical Considerations. Am J Clin Oncol. 2018 Jun;41(6):568-575. doi: 10.1097/COC.0000000000000329. PMID 27635623